CLINICAL TRIAL: NCT02151019
Title: Randomised Phase II Study of Pre-operative 3-D Conformal Radiotherapy (3-DCRT) Versus Intensity Modulated Radiotherapy (IMRT) for Locally Advanced Rectal Cancer
Brief Title: Pre-operative 3-DCRT vs IMRT for Locally Advanced Rectal Cancer
Acronym: TRI-LARC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to futility
Sponsor: Cancer Trials Ireland (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE (ICORG) 12-38
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced Rectal Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Arm (Experimental): 50.4 Gy / 28# external beam pelvic radiotherapy delivered using IMRT
  Interventions: Radiation: IMRT
- Control Arm (No Intervention): 50.4 Gy / 28# external beam pelvic radiotherapy delivered using a 3-Dimensional (3-D) planned technique

INTERVENTIONS:
Radiation: IMRT — IMRT will be given to some patients to enable comparison of the acute grade 2 GI toxicities compared to those patients receiving their radiotherapy by 3-DCRT
  Arms: Experimental Arm

SUMMARY:
The study aims to compare the incidence of acute grade 2 GI toxicity in the Control 3-D Conformal Radiotherapy compared to the Intensity Modulated Radiotherapy (IMRT) arm for locally advanced rectal cancer.

DETAILED DESCRIPTION:
Pre-operative radiotherapy (RT) or chemo-radiotherapy (CRT) is internationally accepted as standard practice in the management of locally advanced rectal cancer.

Multiple randomised trials have proved pre-operative CRT and RT, compared to surgery alone, reduce local recurrence, even prior to optimal surgery, and may improve survival for T3 circumferential resection margin (CRM) negative patients.

This study aims to determine if 3-DCRT or IMRT result in lower incidence of grade 2 GI toxicities.

Acute toxicities will be assessed weekly during radiotherapy, and at 2 and 4 week post treatment.

Late toxicities will be assessed at 3, 6, 9, 12, 18, 24 months post treatment, and annually to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pre-operative pelvic chemo-radiotherapy for histologically confirmed rectal adenocarcinoma, with the following staging: cT3N0-2, cT4N0-2, cT(any)N1-2, cT(any)N(any) CRM at-risk [AJCC version V]
* Staging / imaging of pelvis with MRI, and CT Thorax/Abdomen
* No evidence of metastatic disease
* ECOG Performance Status 0 - 2
* Age > or equal to 18 years
* Provision of written informed consent in line with ICH-GCP guidelines

Exclusion Criteria:

* Previous radiotherapy to the pelvic region
* Patients in whom induction chemotherapy has been delivered prior to chemo- radiotherapy
* History of inflammatory bowel disease
* Previous hip replacement
* Previous bowel surgery (excluding procedures/operations which would not result in small bowel adhesions - at the discretion of the Principal Investigator)
* Patients with other syndromes/conditions associated with increased radiosensitivity
* Any other co-existing malignancies within the past 5 years other than non- melanoma skin cancer
* Pregnancy or lactation at the time of proposed randomisation
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study or if it is felt by the research / medical team that the patient may not be able to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2014-10-17 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Reduction in incidence of grade 2 or higher GI toxicity | 10 years
  To determine if there is a reduction in the incidence of grade 2 or higher acute GI toxicity in the IMRT arm, as compared to the Control / 3-D arm, graded by the NCI-CTCAE Version 4

SECONDARY OUTCOMES:
Compare incidence of acute grade > 2 GU toxicity | 10 years
  To compare the incidence of acute grade > 2 GU toxicity in the IMRT arm, as compared to the Control / 3-D arm, graded by the NCI-CTCAE Version 4
Evaluate incidence of late GI and GU toxicity | 10 years
  To evaluate the incidence of late GI and GU toxicity graded by the NCI-CTCAE Version 4
Rate of loco-regional control | 10 years
  To estimate the rate of loco-regional control by assessing CT / MRI imaging / biopsy
Assess quality of life | 10 years
  To assess QoL according to the EORTC QLQ-C30 and EORTC QLQ-CR29
Rate of disease free survival | 10 years
  To estimate the rate of disease-free survival
Estimate overall survival | 10 years
  To estimate the overall survival rate
Differences in the toxicity profile between the two types of neoadjuvant concomitant chemotherapy, graded by the NCI-CTCAE Version 4 | 10 years
  To compare the differences in the toxicity profile between the two types of neoadjuvant concomitant chemotherapy, graded by the NCI-CTCAE Version 4

CONTACTS AND LOCATIONS:
Overall Officials: Dr Brian O'Neill, MD, Principal Investigator — St Luke's Centre for Radiation Oncology
Locations (3):
- Ireland (3):
  - St Luke's Radiation Oncology Network at Beaumont Hospital, Dublin
  - St Luke's Centre for Radiation Oncology at St James Hospital, Dublin
  - St Luke's Centre for Radiation Oncology at St Lukes Hospital, Dublin